CLINICAL TRIAL: NCT07244471
Title: Water-injecting Endoscopic Submucosal Dissection for Early Gastric Cancer: a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Yingjie Ji, Medical Doctor of Division of Endoscopy Center, Department of Gastroenterology of Shanghai East Hospital, Shanghai East Hospital
Other Study IDs: 20250612IIT0068
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-06

CONDITIONS: Endoscopic Resection; Early Gastric Cancer
Keywords: Endoscopic resection; Early gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Water-injecting ESD: A new ESD method using continuous low-pressure water injection at 1-2 atmosphere with a tip-injected electric knife while dissection simultaneous cutting, dissection, electrocoagulation, and hemostasis, which was so called as water-injecting ESD (W-ESD).
- Conventional ESD: A traditional ESD model. Submucosal injection is performed separately from circumferential cutting, dissection, electrocoagulation, and hemostasis. During the submucosal dissection procedures, submucosal injection is performed with the tip of the knife first, followed by the above operations, rather than simultaneously.

SUMMARY:
Endoscopic submucosal dissection (ESD) is a technically difficult and time-consuming procedure. Several water-jet knives have been developed to address this issue. The aim of this study was to develop a new ESD method using continuous low-pressure water injection at 1-2 atmosphere with a tip-injected electric knife while dissection simultaneous cutting, dissection, electrocoagulation, and hemostasis, which was so called as water-injecting ESD (W-ESD) to treat early gastric cancer and compare the efficacy and safety with conventional methods.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. histologically proven early gastric adenocarcinoma;
3. meeting the absolute or expanded indication for ESD according to the Japanese gastric cancer treatment guidelines 2021 ;
4. Eastern Cooperative Oncology Group performance status ≤ 2;
5. adequate hematological function (hemoglobin ≥ 9 g/dL, platelets ≥ 50 000/mm3，international normalized ratio<1.5);
6. sufficient renal function (serum creatinine ≤ 2.0 mg/dL); and (7) adequate hepatic function (serum aspartate aminotransferase ≤ 100 IU/L, serum alanine aminotransferase ≤ 100 IU/L).

Exclusion Criteria:

1. pregnancy or breastfeeding;
2. difficulty obtaining consent due to psychiatric disorder;
3. multiple lesions;
4. history of gastrectomy or gastrointestinal reconstruction surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who underwent ESD for EGC were enrolled at Shanghai East Hospital between January 2019 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 548 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Total procedure time | Immediately after surgery
  Average time to complete endoscopic resection
Circumferential incision time | Immediately after surgery
  Average time for APC labeling of the lesion margin during circumferential incision
Dissection time | Immediately after surgery
  Average time to complete endoscopic dissection
Dissection speed | Immediately after surgery
  Average speed of endoscopic dissection

SECONDARY OUTCOMES:
Completeness of en bloc resection | Immediately after surgery
  Number of patients with complete lesion resection / Total number of subjects
Adverse event rate | Immediately after surgery and one month post-surgery
  The proportion of adverse events occurring in subjects following surgery (though not necessarily causally related to treatment), encompassing perforation complications, myomere injuries, intraoperative blood loss, thermocoagulation forceps replacements, delayed bleeding, and delayed perforation.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No